CLINICAL TRIAL: NCT02276235
Title: The Therapeutic Effect of Catgut Embedding in Obesity-A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: The Therapeutic Effect of Catgut Embedding in Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, chief medical officer, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101XDAA00024
Record Dates: First submitted 2014-10-14; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Obese Women
Keywords: catgut embedding; obese women; obesity-related hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- catgut embedding group (Experimental): Catgut will be embedding in acupoints as below. Acupoints: Qihai (REN-6), Shuifen (REN-9), bilateral Shuidao (ST-28),bilateral Siman (K-14) ,zusanli(ST-26) Frequency: one time per week Duration: 6 weeks
  Interventions: Device: Catgut embedding group
- sham catgut embedding group (Sham Comparator): The stainless-steel acupuncture needles (3.8cm long) was inserted into 23 gouge needle as plunger without chromic catgut in front of the syringe needle. All the procedure will be performed as in catgut embedding group.
  Acupoints: Qihai (REN-6), Shuifen (REN-9), bilateral Shuidao (ST-28),bilateral Siman (K-14) ,zusanli(ST-26)
  The other procedure were the same as catgut embedding group Frequency: one time per week Duration: 6 weeks
  Interventions: Device: sham catgut embedding group

INTERVENTIONS:
Device: Catgut embedding group — An extensive form of acupuncture that involves weekly infixing self-absorptive chromic catgut sutures into acupoints with a specialised needle under antiseptic precautions. The catgut then stimulate those points over a long period. The stainless-steel acupuncture needles (3.8cm long) was inserted into 23 gouge needle as plunger with chromic catgut in front of the syringe needle. Catgut will be embedding in acupoints as below.
  Acupoints: Qihai (REN-6), Shuifen (REN-9), bilateral Shuidao (ST-28),bilateral Siman (K-14) ,zusanli(ST-26)
  Other Names: acupoint catgut embedding
  Arms: catgut embedding group
Device: sham catgut embedding group — The stainless-steel acupuncture needles (3.8cm long) was inserted into 23 gouge needle as plunger without chromic catgut in front of the syringe needle. Catgut will be embedding in acupoints as below.
  Acupoints: Qihai (REN-6), Shuifen (REN-9), bilateral Shuidao (ST-28),bilateral Siman (K-14) ,zusanli(ST-26)
  Other Names: sham acupoint catgut embedding
  Arms: sham catgut embedding group

SUMMARY:
The aim of this double-blind, randomized, placebo-controlled trial is to evaluate the therapeutic effects of acupoint stimulation by catgut embedding on complexion, quality of life, lipid profile, inflammatory markers, and obesity-related hormone peptide of obese women.

DETAILED DESCRIPTION:
We will recruit 90 females aged from 16 year-old to 65 year-old with body mass index(BMI) 27㎞/㎡ and waist circumference≧80cm. After inform consent, they will be randomly assigned into two groups. In group A, catgut embedding will be applied to six acupuncture points on the abdomen including Qihai (Ren-6), Shuifen (REN-9), bilateral shuidao (ST-28) and Siman (ST-26), which have been proved to be effective on obesity in our previous study, once each week for six times. In group B, sham catgut embedding will be applied on the same acupoints once each week for six weeks. This trial will go on for six weeks with six course of treatment.

Our primary outcome measurements is complexion which included body mass index(BMI),waist circumstances, and waist-hip ratio. In our second outcome measurments, we will evaluate the life quality of these patients using 12-Item Short Form Health Survey (SF-12) which developed for the Medical Outcomes Study (MOS) and also using questionnaire of quality of life that was designated by World Health Organization. We will also classify the patients by questionnaire designed for TCM syndrome of obesity. We will check blood test included lipid profile (TG, Chol, HDL-C, LDL-C), inflammatory markers, and hormone peptide related to obesity such as insulin,leptin,ghrelin,adiponectin. Each enrolling patients will be evaluated at the baseline before treatment and after 6 times treatments completed by above parameters to find out the therapeutic effects and mechanism of catgut embedding in acupoints in obese women.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) ≥ 27 kg/m2 waist circumference (WC) ≥ 80 cm and willing to participate in and fill out the questionnaires for this trial.

Exclusion Criteria:

* Endocrine disease(Thyroid disease, pituitary disease, diabetes mellitus) Autoimmune disease（SLE、SSS、RA） Heart disease(Heart failure, arrhythmia etc.） Abnormal liver function（GOT>80U/L、GPT>80U/L） Abnormal kidney function（serum creatinine>2.5 mg/dL） Stroke disease in past one year Under breast feeding or pregnancy Coagulation disorder Subjects with keloid disorder Accept weight reduction treatment in last two months

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
body weight | assessed at each time before procedures and one week after the 6th treatment, an expected average of 7 weeks
body mass index | assessed at each time before procedures and one week after the 6th treatment, an expected average of 7 weeks
waist circumference | assessed at each time before procedures and one week after the 6th treatment, an expected average of 7 weeks
hip circumference | assessed at each time before procedures and one week after the 6th treatment, an expected average of 7 weeks

SECONDARY OUTCOMES:
cholesterol | Assess at baseline and after 6 weeks of treatment
  cholesterol (Chol),
triglyceride (TG) | Assess at baseline and after 6 weeks of treatment
  triglyceride (TG),
low-density lipoprotein cholesterol (LDL-C) | Assess at baseline and after 6 weeks of treatment
  low-density lipoprotein cholesterol (LDL-C)
High-density lipoprotein cholesterol(HDL-C) | Assess at baseline and after 6 weeks of treatment
  High-density lipoprotein cholesterol(HDL-C)
Quality of life | Assess at baseline and after 6 weeks of treatment
  short-form 12 items and WHOQOLBREF
Questionnaire on traditional Chinese medicine syndrome groups | Assess at baseline and after 6 weeks of treatment
  Obesity subjects will be classified into six groups including stomach heat, yin deficiency, qi stagnation, qi deficiency, kidney deficiency and blood stasis With more than two "yes"in items, patient will be classified to that kind of syndrome
sugar | Assess at baseline and after 6 weeks of treatment
  AC sugar,
glycohemoglobin | Assess at baseline and after 6 weeks of treatment
  glycohemoglobin (HbA1c),
liver function | Assess at baseline and after 6 weeks of treatment
  ALT
kidney function | Assess at baseline and after 6 weeks of treatment
  Cr
inflammatory markers | Assess at baseline and after 6 weeks of treatment
  hsCRP

CONTACTS AND LOCATIONS:
Locations (1):
- Branch of Chinese Medicine, Taipei City Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Result] Huang CY, Choong MY, Li TS. Treatment of obesity by catgut embedding: an evidence-based systematic analysis. Acupunct Med. 2012 Sep;30(3):233-4. doi: 10.1136/acupmed-2012-010176. Epub 2012 Jul 7. No abstract available. PMID 22773366
- [Result] Liao JQ, Song X, Chen Y, Liang LC, Wang SX. [Clinical randomized controlled trials of acupoint catgut-embedding for simple obesity: a meta-analysis]. Zhongguo Zhen Jiu. 2014 Jun;34(6):621-6. Chinese. PMID 25112111